CLINICAL TRIAL: NCT01230879
Title: Study of Bronchoalveolar Lung Remodeling in Subjects From 60 Years Free of Progressive Lung Disease: Structure-function Analysis
Brief Title: Effect of Ageing on Airway Remodeling
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8268
Record Dates: First submitted 2010-08-04; First posted 2010-10-29 (Estimated); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Aging
Keywords: Aging lung; Airway remodeling; Airway segmentation; Chest CT
MeSH Terms: conditions — Airway Remodeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 60 - 70 years old (Experimental): EFR and TDM
  Interventions: Other: EFR and TDM
- 71 - 80 years old (Experimental): EFR and TDM
  Interventions: Other: EFR and TDM
- 81 - 95 years old (Experimental): EFR and TDM
  Interventions: Other: EFR and TDM

INTERVENTIONS:
Other: EFR and TDM — EFR : Pulmonary function test TDM : tomodensitometry

SUMMARY:
The aim of the study is to investigate the relationship between aging and morphological changes in the lung. 120 consecutive healthy volunteers over 60 years will be enrolled for this trial.

DETAILED DESCRIPTION:
Chest multidetector CT without injection and spirometry data will be obtained from a multicentric sample of individuals between 60 and 95 years of ageExclusion criteria were current smoking, history of smoking within the past 10 years, any known chronic or acute pulmonary disease. Individuals treated with Amiodarone, Bleomycin or methotrexate were excludedOutcome

ELIGIBILITY:
Inclusion Criteria:

* People from 60 to 95 years old free from chest disease or history of chest disease

Exclusion Criteria:

* Chronic cough
* Dyspnea
* Sinonasal or chest infection during enrollment
* Myocardial infarction.
* Current smoker or past smoker with more than 10 pack year intoxication

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2009-07-15; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Bronchial wall thickness | 1 day
  Bronchial wall thickness and remodeling associated with aging

CONTACTS AND LOCATIONS:
Overall Officials: BOMMART Sebastien, MD, Principal Investigator — University Montpellier Hospital
Locations (1):
- University Montpellier Hospital, Montpellier, France

REFERENCES:
- [Result] Bommart S, Marin G, Bourdin A, Molinari N, Klein F, Hayot M, Vachier I, Chanez P, Mercier J, Vernhet-Kovacsik H. Relationship between CT air trapping criteria and lung function in small airway impairment quantification. BMC Pulm Med. 2014 Feb 28;14:29. doi: 10.1186/1471-2466-14-29. PMID 24581147